CLINICAL TRIAL: NCT04972084
Title: Three-dimensional Evaluation of the Efficacy of Powerscope Appliance in Treatment of Skeletal Class 2 Malocclusion: A Prospective Clinical Study
Brief Title: 3D Evaluation of Powerscope Appliance in Treatment of Skeletal Class 2 Malocclusion
Acronym: Powerscope app
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hany Essam Mohamed El-Hossainy, Master's degree candidate, Orthodontic department, Al-Azhar University, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3D Powerscope Class II ttt
Record Dates: First submitted 2021-07-01; First posted 2021-07-22 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Class II Malocclusion, Division 1
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Powerscope group (Experimental): Class II patients which will receive treatment using Powerscope appliance
  Interventions: Device: Powerscope group

INTERVENTIONS:
Device: Powerscope group — Treatment of Class II malocclusions using Powerscope appliance

SUMMARY:
The study is aiming to evaluate the efficacy of Powerscope appliance in treatment of skeletal Class 2 malocclusion by three-dimensional image. Powerscope appliance is a hybrid fixed functional appliance used for treatment of Class II malocclusion with a retruded mandible.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy post pubertal female patients of age range 14 to 16 years old, manifesting features of post pubertal cervical vertebrae maturational stages 4, 5 and 6 (deceleration, maturation, and completion).
2. Skeletal class 2 malocclusion of ANB angle greater than 4° with retrognathic mandible.
3. Class II division 1 malocclusion with at least an end-on Class II molar relationship.
4. Presence of all permanent dentition excluding third molars.
5. Good oral hygiene.

Exclusion Criteria:

1. History of previous orthodontic treatment.
2. Any systemic disease that could affect the orthodontic treatment.
3. Patients with periodontal diseases.
4. Patients with temporomandibular disorders.

Ages: 14 Years to 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Only females are enrolled in the study
Enrollment: 12 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-09-05 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
The Condylar head volumetric changes | six months
  The change in Condylar head volume before and after usage of Powerscope appliance

SECONDARY OUTCOMES:
Mandibular length | six months
  The change in the length of the mandible

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar university, Faculty of oral and dental medicine, Cairo, Naser City, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: A year